#### RESEARCH PROTOCOL

**Study Number:** Title: A Randomized, Double Blind, Placebo-Controlled Single Center Phase 2 Pilot Study to Assess the Safety and Efficacy of Off-label Subcutaneous Administration of Erenumab-aooe in Patients with Temporomandibular Disorder Sponsor: Indiana University\* **Investigation Site:** Oral Health Research Institute Indiana University School of Dentistry **Principal Investigator:** Domenick T. Zero, DDS, MS, Oral Health Research Institute 415 Lansing Street Indianapolis, IN 46202-2876 Phone: 317-274-8822 FAX: 317-274-5425 Email: dzero@iu.edu **Co-Principal Investigator:** Harold C. Avila, DDS, MS Adjunct Clinical Assistant Professor Department of Oral Pathology, Medicine and Radiology Indiana University School of Dentistry **Co-Investigator:** Kurt Kroenke, MD, MACP Chancellor's Professor, IUPUI General Internal Medicine Indiana University Center for Health Services/Outcomes Research, Regenstrief Institute 1101 W. 10th Street Indianapolis, IN 46202 **Study Dentist** Ana Gossweiler, DDS, MSD Oral Health Research Institute Statistician: George Eckert, MAS Department of Biostatistics Indiana University School of Medicine Study Manager: **TBD** Version: Final: Revised 01FEB2021

Amendment 8: January 12, 2023

<sup>\*</sup> Funded by Amgen through Investigator Sponsored Studies (ISS) Program (CAMG334AUS01T)

# **Table of Contents**

| List of | Abbreviations | 3 |
|---|---|---|
| 1. B | ackground & Rationale | 4 |
| 2. S | tudy Objectives and Outcome Measures | 5 |
| 2.1 | Primary Objective and Outcome Measure | 5 |
| 2.2 | Secondary Objective and Outcome Measures | 5 |
| 3. S | tudy Design | 5 |
| 4. S | tudy Population | 6 |
| 4.1 | Inclusion Criteria | 6 |
| 4.2 | Exclusion Criteria | 6 |
| 4.3 | Enrollment Procedures | 7 |
| 5. T | reatments | 8 |
| 5.1 | Study Treatments | 8 |
| 5.2 | Treatment Arms | 8 |
| 5.3 | Treatment assignment and randomization | 8 |
| 5.4 | Treatment blinding | 8 |
| 5.5 | Dispensing of study drug | 8 |
| 6. V | isit Schedule and Assessments | 9 |
| 7. S | afety Monitoring | 11 |
| 7.1 | Adverse Events | 11 |
| 7.2 | Serious Adverse Events | |
| 7.3 | Study Withdrawal/Discontinuation | |
| 8. D | ata Analysis | 12 |
| 8.1 | Sample size calculations | |
| 9. R | leferences | |
| 10. | Appendices | |
| | endix A – TMD Symptoms | |
| App | endix B – TMD Treatments | 16 |
| App | endix C – Diagnostic Criteria for Temporomandibular Disorders Symptom Question | |
| | endix D – Brief Pain Inventory (BPI) | |
| | endix E – PEG (Pain, Enjoyment, General Activity) Scale and Pain Medication | 20 |
| | essmentenjoyment, General Activity) Scale and Fain Medication | 22 |
| | endix F – Patient Global Impression of Change (PGIC) | |
| • • • | endix G – Jaw Function Limitation Scale (JFLS-8) | |
| | endix H – Depressive and anxiety symptoms (PHQ-4) | |
| | endix I – Somatic symptom severity as measured by the SSS-8 | |
| 11. | Table 1 | |

# **List of Abbreviations**

| AE | Adverse Event |
|---|---|
| BPI | Brief Pain Inventory |
| CFR | Code of Federal Regulations |
| CGRP | Calcitonin Gene Related Peptide |
| CM | Chronic Migraine |
| COPCs | Chronic Overlapping Pain Conditions COPCs |
| CPAP | Continuous Positive Airway Pressure |
| CRF | Case Report Form |
| DC/TMD | Diagnostic Criteria/Temporomandibular Disorder |
| EREN | Erenumab-aooe |
| EREN-P | Placebo |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| IRB | Institutional Review Board |
| IUPUI | Indiana University Purdue University Indianapolis |
| IUSD | Indiana University School of Dentistry |
| JFLS | Jaw Function Limitation Scale |
| NIH/NIDCR | National Institutes of Health/National Institutes of Dental and Craniofacial Research |
| PEG | Pain, Enjoyment, General Activity Scale |
| PGIC | Patient Global Impression of Change |
| PHQ-4 | Patient Health Questionnaire |
| PI | Principal Investigator |
| SAE | Serious Adverse Event |
| S.C. | Subcutaneous |
| SOP | Standard Operating Procedure |
| SSS-8 | Somatic Symptom Scale |
| TGV | Trigeminovascular Pathway |
| TMD | Temporomandibular Disorder |
| UmMa(s) | Human Monoclonal Antibody(s) |

# 1. Background & Rationale

Aimovig® [erenumab (EREN)] is a first in class FDA-approved human monoclonal antibody (UmAb) for the prevention of migraine in adults. It selectively targets and blocks the calcitonin gene-related peptide (CGRP) receptor, disrupting a key component of migraine pathophysiology (Hargreaves & Olesen, 2019). Several studies have provided evidence of the safety and efficacy of Aimovig® in reducing the frequency of migraine compared to placebo (Goadsby et al., 2017; Tepper et al., 2017). Furthermore, an open-label longer-term study found that Aimovig® was safe and well-tolerated with a safety profile consistent with shorter-term placebo-controlled studies (Ashina et al., 2020), through 5-years of treatment. Aimovig® has rapidly become a widely accepted prescription drug for the prevention of migraines, including episodic migraine and chronic migraine (CM) along with other anti-CGRP monoclonal antibody-based therapies (Yuan et al., 2019).

Temporomandibular Disorders (TMD) are known to be co-morbid with the medical diagnosis of CM (Speciali, 2015). TMD symptoms are numerous and chronic in nature (see appendix A) and TMD treatments are more numerous than symptoms and are predictable only in their unpredictability (see Appendix B). Most patients experiencing TMD find it to be a chronic, untreatable condition. In the US alone, TMDs are the second most commonly occurring musculoskeletal conditions resulting in pain and disability (after chronic low back pain), affecting approximately 5 to 12% of the population, with an annual cost estimated at \$4 billion (NIH/NIDCR). There is increasing interest in the concept of Chronic Overlapping Pain Conditions (COPCs), which include TMD, fibromyalgia, irritable bowel syndrome, vulvodynia, myalgic encephalomyelitis/chronic fatigue syndrome, interstitial cystitis/painful bladder syndrome, endometriosis, chronic tension-type headache, migraine headache, and chronic lower back pain that may have common biopsychosocial factors (Maixner et al., 2016).

Co-Principal Investigator, Dr. Harold C. Avila, has treated several patients that presented with chronic TMD pain and a history of migraines headaches, which have responded positively to off-label administration of Aimovig®. Anecdotally, five of Dr. Avila's TMD patients were treated with Aimovig® along with his standard therapy. Of these, three patients experienced substantial life-changing relief of TMD pain symptoms. Another patient initially experienced substantial pain relief, which declined slightly over two months. The last patient stopped taking Aimovig® due to elevated blood pressure, which is not an adverse event associated with Aimovig® in the published clinical trials (Goadsby et al., 2017; Tepper et al., 2017); however, the development of hypertension and worsening of pre-existing hypertension have been reported following the use of AIMOVIG in the postmarketing setting (FDA-approved Patient Labeling).

CM is thought to originate within the trigeminovascular pathway (TGV) (Noseda & Burstein, 2013). TMD is also considered to originate within the TGV (de Leeuw, 2018). Thus, our working hypothesis is that a CGRP receptor antagonist for treatment of CM will also be effective in reducing TMD pain and related symptoms. To test this hypothesis, we applied several validated measures: Brief Pain Inventory (BPI) (Kean et al., 2016); PEG (Pain, Enjoyment, General Activity) Scale (Krebs et al., 2009); an assessment of daily pain medication; Patient Global Impression of Change (PGIC) (Kroenke et al., 2018); Jaw Function Limitation Scale (JFLS) (Ohrbach et al., 2008); Patient Health Questionnaire (PHQ-4) (Kroenke et al., 2009); and Somatic Symptom Scale (SSS-8) (Toussaint et al., 2017).

The purpose of this proof of concept study was to evaluate the safety and efficacy of the off-label use of Aimovig® (EREN) in reducing Temporomandibular Disorder (TMD) pain compared to placebo.

# 2. Study Objectives and Outcome Measures

#### 2.1 Primary Objective and Outcome Measure

To assess the effects of Aimovig® (EREN) compared to placebo (EREN-P) based on the change in mean between-group difference in pain using the Brief Pain Inventory (BPI) 4-item pain severity/intensity scale during the 20-week trial. The BPI is a validated and widely used outcome measures in chronic pain trials (Kean et al., 2016; Kroenke et al., 2019). We postulated that Aimovig® will be superior to placebo in reducing pain intensity/severity over 20 weeks.

### 2.2 Secondary Objective and Outcome Measures

To assess the effects of Aimovig® (EREN) compared to placebo (EREN-P) based on the change in mean between-group difference in secondary outcomes during the 20-week trial and after 24 weeks (two months after the last treatment). The outcome measures are based on consensus recommendations for research assessments in chronic pain and TMD research (Ohrbach et al., 2016; Kroenke et al., 2019). We postulated that Aimovig® will be superior to placebo in improving several secondary outcomes including:

- a) Pain interference as measured by the BPI interference scale
- b) Trajectory of pain improvement based on changes in daily reporting of pain using the PEG (Pain, Enjoyment, General Activity) Scale as measured using an app downloaded on the subject's smartphone or for individuals without smartphones at baseline and every 4 weeks over the 24-week study period
- c) Days of use of TMD pain-specific medication per month
- d) Global improvement in pain as measured by the Patient Global Impression of Change (PGIC)
- e) Jaw function as measured by the Jaw Function Limitation Scale (JFLS-8)
- f) Depressive and anxiety symptoms as measured by the Patient Health Questionnaire (PHQ-4)
- g) Somatic symptom severity as measured by the Somatic Symptoms Scale (SSS-8)
- h) Safety and tolerance as measured by incidence of AEs and SAEs

#### 3. Study Design

This was a 24-week, randomized, double-blinded, placebo-controlled, parallel group proof-of-concept study with two arms (active and placebo). The plan was to enroll 30 subjects. There was a four-week screening period to identify subjects that meet the diagnostic criteria (DC/TMD) for "myalgia", recommended by the International RDC/TMD Consortium Network and Orofacial Pain Special Interest Group (Schiffman et al., 2014). The Diagnostic Criteria for Temporomandibular Disorders Symptom Questionnaire and DC/TMD Examination Form (Ohrbach, 2016) was used during Screening and Baseline visits to confirm the TMD diagnosis and determine whether subjects met the inclusion/exclusion criteria.

Subjects attended a Screening visit followed by Baseline visit to randomize eligible subjects to active (EREN) or placebo (EREN-P). During the Baseline visit and Wks 4, 8, 12, and 16, subjects received treatment with either 140 mg of EREN or Placebo administered by subcutaneous injection. At Baseline and Wks 4, 8, 12, 16, 20, and 24 subjects were instructed to complete the Brief Pain Inventory (BPI) (Kean et al., 2016); PEG (Pain, Enjoyment, General Activity) Scale (Krebs et al., 2009); pain mediation assessment; Patient Global Impression of Change (PGIC)

(Kroenke et al., 2018) (except for Baseline visit); Jaw Function Limitation Scale (JFLS) (Ohrbach et al., 2008); Patient Health Questionnaire (PHQ-4) (Kroenke et al., 2009); and Somatic Symptom Scale (SSS-8) (Toussaint et al., 2017). These visits also included review of continuance criteria and adverse event collection.

At the Screening and Baseline visits the subjects were instructed on how to use the PEG Scale and pain use assessment app, which was downloaded on their smartphone, to provide a daily assessment of their pain intensity and interference with enjoyment and general activity (PEG) and their daily used of pain medications. Subjects who did not own a smartphone or were unwilling to use the app on a daily basis only completed the PEG and pain medication assessment at the Baseline visit and all subsequent visits using the app onsite.

# 4. Study Population

The study population consisted of male and female subjects diagnosed as having pain-related TMD using the diagnostic criteria (DC/TMD) for "myalgia", recommended by the International RDC/TMD Consortium Network and Orofacial Pain Special Interest Group (Schiffman et al., 2014). The goal was to recruit 30 subjects that fulfill the inclusion and exclusion criteria. It was anticipated that 24 subjects (12 in each treatment group) will complete all aspects of the study.

#### 4.1 Inclusion Criteria

Subjects eligible for inclusion in the study must have met all of the following criteria:

- 1. Signed the informed consent;
- 2. Have a history of head, face, neck and/or shoulder pain for longer than 3 months;
- Have a diagnosis of myalgia based on clinical examination using DC/TMD criteria;
- 4. Age 18 years and younger than 60 years;
- 5. Have a good knowledge of the English language;
- 6. Able to understand and comply with the study requirements; and
- 7. If taking prescription pain medications, the dose regimen must be stable for at least 2 months prior to the screening visit.

#### 4.2 Exclusion Criteria

Subjects that met any of the following criteria were not eligible for inclusion:

- 1. Lacking stable bilateral posterior occlusion;
- 2. Currently uses a complete maxillary or mandibular prosthetic denture;
- 3. Currently pregnant or plan to become pregnant;
- 4. Breastfeeding or plan to breastfeed;
- 5. Allergic to erenumab-aooe or any of the ingredients in Aimovig® (acetate, polysorbate 80, and sucrose);
- 6. Allergic to rubber or latex;
- 7. Currently undergoing TMD treatment elsewhere. Exception: patients undergoing TMD treatment involving the use of oral orthotics for a minimum of 3 months prior to Screening can be considered eligible for the study;

- 8. Started orthodontic treatment during the 3 months prior to Screening;
- 9. Currently included in other experimental protocols within the last 30 days or 5 half-lives before enrollment;
- 10. Having 8 or more migraine days during the past 4 weeks;
- 11. Started receiving massage, acupuncture or physical therapy treatment of the head, neck or shoulders during the previous 3 months prior to Screening;
- 12. History of unstable or acute severe non-head, neck or shoulder pain;
- 13. History of traumatic brain injury;
- 14. History of surgical treatment or recommended surgical treatment for TMD;
- 15. History of ongoing, unresolved disability litigation;
- 16. History of drug abuse;
- 17. Started treatment for moderate to severe sleep apnea requiring CPAP or oral mandibular repositioning appliance during the previous 3 months prior to Screening;
- 18. Anything that would place the subjects at increased risk or preclude the individual's full compliance with or completion of the study (e.g., medical condition, laboratory finding, physical exam finding logistical complication);
- 19. History of previously receiving erenumab-aooe or other anti-CGRP pathway therapies, including anti-CGRP and anti-CGRP receptor monoclonal antibodies and small molecule CGRP receptor antagonists (gepants);
- 20. History of chronic constipation and/or using medication associated with decreased gastrointestinal motility; and
- 21. History of uncontrolled hypertension or risk factors for hypertension.

#### 4.3 Enrollment Procedures

Subjects were recruited using fliers and advertisements placed in the Indiana University (IU) School of Dentistry (IUSD) and other locations on the Indiana University Purdue University Indianapolis (IUPUI) campus including IU Health facilities. Fliers may also be posted on Facebook.

Dr. Avila may send approved study information to persons who may have TMD and he may also mention the study during planned radio interviews about TMD. Dr. Avila's website will not mention research.

Persons responding to an advertisement will be given a brief description of the study and asked a series of questions related to the inclusion/exclusion criteria using an IRB approved phone script. Those who are interested and appear to meet the study requirements will be scheduled for a screening visit at the Oral Health Research Institute (OHRI).

Additionally, contact information was obtained from Regenstrief for IU Health patients who have indicated they have TMJ problems and are willing to be contacted for future studies. Once contact information was obtained, the OH study coordinator contacted the potential subjects by telephone to see if they were interested in attending a screening visit.

#### 5. Treatments

#### 5.1 Study Treatments

Investigational drug: erenumab-aooe (EREN) 140 mg, for s.c. injections, provided by Amgen

**Placebo**: liquid placebo (EREN-P), for s.c. injections provided by Amgen

Amgen provided the active and placebo free of charge through the Investigator Sponsored Studies (ISS) Program (CAMG334AUS01T).

#### 5.2 Treatment Arms

Subjects were assigned at baseline to one of the two treatment arms:

- Arm A: erenumab-aooe (EREN) 140 mg s.c. administered every four weeks for a total of five treatments
- Arm B: placebo (EREN-P) s.c. administered every four weeks for a total of five treatments

#### 5.3 Treatment assignment and randomization

Subjects were randomized and stratified based on gender into two groups using block randomization based on a schedule provided by the study statistician, George Eckert, Indiana University School of Medicine Department of Biostatistics.

The randomization code was provided to Amgen as part of the ISS contract agreement.

#### 5.4 Treatment blinding

Subjects, investigators and study staff will remain blind to the identity of the treatment from the time of randomization until database lock. The randomization code will be kept strictly confidential and the identity of the study drug treatments will be concealed using identical packaging and labeling. The blind will only be broken in an emergency where it is essential to know which treatment a subject received in order to give the appropriate medical care.

#### 5.5 Dispensing of study drug

The investigational products (EREN and EREN-P) supplied in prefilled syringes will be shipped by Amgen to the attention of the unblinded IU Health Investigational Drug Services Pharmacy. The IU Health Pharmacy will dispense the investigational products according to a randomization schedule provided by the study statistician, George Eckert. A written prescription order form will be completed by the licensed study dentist and submitted to the pharmacy each time study drug is requested for a subject. Doses will be administered in the upper arm, thigh, or abdomen by a study dentist qualified in s.c. drug administration.

Study product will be stored and handled according to labeling instructions: store refrigerated at 2°C to 8°C (36°F to 46°F) in the original carton to protect from light until time of use; do not freeze; and do not shake; leave the prefilled syringe at room temperature for at least 30 minutes before injecting. The investigational products will be stored in a secured area of the IU Health Investigation Drug Services Pharmacy to which only the pharmacy staff have access.

The IU Health pharmacy will maintain adequate records documenting the receipt, use, loss, or other disposition of the products on the electronic Investigational Agent Accountability Record. The log will identify the products and account for the disposition including specific dates and

quantities used/dispensed and returned, as applicable. The log will capture the electronic signatures of the site designees who dispensed and verified the products.

The clinical site, OHRI, working with the pharmacy will also maintain a Drug Administration Form documenting the date and time of transport to the blinded site staff, the date and signature of the blinded site staff receiving the study drug, the date and time the study drug was received from the pharmacy, the date and time the study drug was administered, and the injection site body location.

#### 6. Visit Schedule and Assessments

#### **Study Schedule**

| Period | Screening | | Treatment Period | | | | | |
|---|---|---|---|---|---|---|---|---|
| Visit Name | Screening | Baseline | Wk 4 | Wk 8 | Wk 12 | Wk 16 | Wk 20 | Wk 24 |
| Days | -28 to -1 | 1 | 29 | 57 | 85 | 113 | 141 | 169 |
| Weeks | -4 to -1 | 0 | 4 | 8 | 12 | 16 | 20 | 24 |
| Informed consent | X | | | | | | | |
| Randomization | | X | | | | | | |
| Study drug administration | | X | Х | Х | Х | X | | |
| Inclusion / Exclusion criteria | X | | | | | | | |
| Demography | X | | | | | | | |
| Medical history/current medical conditions | X | | | | | | | |
| Prior therapy for TMD | Х | | | | | | | |
| Adverse Events | X | X | Χ | Х | Х | Х | X | Χ |
| Concomitant medications | X | X | Χ | Х | X | X | X | Χ |
| Familiarize with PEG App | X | X | | | | | | |
| BPI, PEG and pain<br>medication assessment<br>(daily), JFLS-8, PHQ-4,<br>SSS-8 | | Х | Х | Х | Х | Х | Х | Х |
| PGIC | | | Χ | Х | Х | Х | X | X |

<u>Screening Visit</u>: Subjects will complete the informed consent process, being given ample time to review the consent and to ask any questions they have before deciding if they wish to participate. Those interested will sign and date their informed consent and the consent will also

be signed and dated by the person reviewing the consent process with them. Subjects will receive a signed copy of their consent before leaving this visit. A Study Dentist qualified to diagnosis TMD will review the potential subject's health history, medications and TMD history for the inclusion and exclusion criteria.

The Diagnostic Criteria for Temporomandibular Disorders Symptom Questionnaire (Appendix C) and DC/TMD Examination Form (Ohrbach, 2016) will be used to confirm the TMD diagnosis and determine whether subjects meet the inclusion/exclusion criteria. To meet the diagnostic criteria for TMD Myalgia (IDC-9 729; ICD-10 M79.1) (Schiffman et al., 2014), subjects must have a history of pain of muscle origin that is affected by jaw movement, function, or parafunction, and demonstrate replication of this pain with provocation testing of the masticatory muscles. The specific criteria (Schiffman et al., 2014) include having a positive history for both pain in the jaw, temple, in the ear, or in front of ear and pain modified with jaw movement, function or parafunction. During clinical examination, subjects must have a confirmation of pain in the temporalis or masseter muscle(s) and report familiar pain in the temporalis or masseter muscle(s) with at least one of the following provocation tests: palpation of the temporalis or masseter muscle(s) or maximum unassisted or assisted opening movement(s).

Subjects with smartphones will be asked to download the MyCap app and will then be trained on completing the PEG Scale and the pain medication assessment questions using their smartphone. The subject will be scheduled to return to the study site for their Baseline visit.

Baseline, Wk 4, 8, 12, and 16 Visits: The subject's medical history, medications and continuance criteria will be reviewed to assure the subject still qualifies to participate in the study. The Diagnostic Criteria for Temporomandibular Disorders Symptom Questionnaire (Appendix C) and DC/TMD Examination Form will be used to confirm the TMD diagnosis and determine whether subjects meet the inclusion/exclusion criteria. In addition, the subjects will be assessed using the Brief Pain Inventory (BPI) (Appendix D), PEG (Pain, Enjoyment, General Activity) Scale and pain medication assessment (Appendix E), Jaw Function Limitation Scale (JFLS) (Appendix G), Patient Health Questionnaire (PHQ-4) (Appendix H), and Somatic Symptom Scale (SSS-8) (Appendix I). Starting at week 4 the subjects will also be assessed using global improvement in pain as measured by the Patient Global Impression of Change (PGIC) (Appendix F).

The subject will receive their assigned treatment (EREN or EREN-P) based on the randomization scheme at baseline and Wk 4, 8, 12, and 16.

The procedure for texting each day will be reviewed with the subject and a practice text will be sent to assure communication is accurate. Subjects without smartphones will only be required complete the PEG Scale and pain medication assessment questions using the app onsite at Baseline and at all subsequent study visits.

Adverse events will be assessed and documented, and the subjects will be schedule for their next visit.

<u>Wk 20 End of Treatment Period Visit</u>: Subjects will be assessed using the BPI, PEG and pain medication assessment (app), PGIC, JFLS, PHQ-4, and SSS-8. Adverse events will be assessed and documented, and the subjects will be schedule for their next visit.

Wk 24 Post-Treatment Follow-up Visit: Subjects will return for follow-up examination and assessed using the BPI, PEG and pain medication assessment (app), PGIC, JFLS, PHQ-4, and SSS-8. Adverse events will be assessed and documented.

# 7. Safety Monitoring

This study will be conducted in compliance with the US Code of Federal Regulations (CRF) governing informed consent (21 CFR 50), Institutional Review Board (IRB) (21 CFR 56), and with applicable regulations governing Investigator conduct (21 CFR 312).

This study will be performed according to GCPs. SOPs for all procedures are on file with the Quality Assurance staff of the Oral Health Research Institute.

All study staff who have direct subject contact will be required to review the WARNINGS AND PRECAUTIONS for Hypersensitivity Reactions, Constipation with Serious Complications and Hypertension found in Section 5 of the US Prescribing Information (USPI) for Aimovig®.

https://www.pi.amgen.com/~/media/amgen/repositorysites/pi-amgen-com/aimovig/aimovig pi hcp english.ashx

#### 7.1 Adverse Events

Subjects will be questioned regarding any general health or oral complaints and symptoms they have experienced during each visit. Any findings will be documented on the AE CRF. In the event of subjects reporting AEs outside the scheduled clinical visit, the Investigator will assess them at the earliest opportunity.

All AEs, regardless of severity or relationship to the treatments, will be recorded. Serious AEs include any events resulting in death, decreased life expectancy, life-threatening situations, persistent or permanent disability/incapacity, hospitalization, or congenital anomaly/birth defect. In addition, other important medical events that are deemed clinically important/serious based on PI judgement will be recorded as AEs. Within 24 hours, the Investigator will submit a written report to Amgen documenting the circumstances of the serious AE.

#### 7.2 Serious Adverse Events

Safety monitoring for this study will focus on adverse events related to treatment use and unanticipated problems involving risks to participants, including unanticipated problems that meet the definition of a serious adverse event. At each visit, subjects will be queried about any adverse events that may have occurred since their last visit, regardless of direct relationship to treatment use. Adverse events will be recorded on an Adverse Event form. Abnormalities, or worsening of pre-existing conditions, observed by the examiner or reported by the subject that occur at any visit will be recorded on the AE CRF. All AEs will be transcribed onto a log, which will be monitored by the PI to determine if the nature, frequency, or severity of an event meets the criteria for prompt reporting. All adverse events will be reported to the IRB during annual review.

The PI will be notified immediately if a serious adverse event occurs. All serious adverse events that meet the prompt reporting requirements will be reported to the IRB within 5 business days. Serious adverse events include: any event resulting in death, is life-threatening, requires hospitalization, results in disability/permanent damage, congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage, and/or other medical events.

The study site will be responsible for reporting SAEs to Amgen in accordance with the Amgen ISS Program contract requirements.

The study site will be responsible for reporting all safety information to Amgen in accordance with their reporting requirements (<u>Table 1</u>).

### 7.3 Study Withdrawal/Discontinuation

Subjects may withdrawal or discontinue from the clinical trial at any time without penalty or loss. Subjects will be advised at the start of the trial that they may withdraw from the trial at any time, without giving a reason. Subjects may be withdrawn by the Principal Investigator for the following reasons:

- the volunteer wishes to withdraw;
- if, in the opinion of the Investigator, it is in the best interests of the subject;
- if serious adverse reactions occur;
- inter-current illness occurs;
- there is a significant violation of the prohibitions and restrictions;
- development of an exclusion criterion.

Withdrawals due to non-attendance must be followed up to attempt to obtain the reason that the subject is 'lost to follow up'. Subjects who are lost to follow up will be encouraged to return to the site for an exit visit. Subjects withdrawn for medical reasons will be referred to a physician /dentist. Their condition will be monitored until it is resolved or clinically non-significant. All withdrawals and the reason for withdrawal will be documented. Withdrawn subjects will not be replaced.

#### 8. Data Analysis

Mixed model repeated measures (MMRM) analysis will be used to evaluate changes over time in the BPI pain severity/intensity scale and BPI total score, PEG Scale total score and daily pain, days of use of pain medication and TMD pain-specific medication per month, JFLS-8, PHQ-4 anxiety and depression, SSS-8 Scale, and PGIC pain change within and between treatment groups. The MMRM will include factors for treatment group, time, and their interaction. Time will be repeated within subject. The MMRM will also include gender as a covariate due to stratification by gender in the randomization. The distribution of the outcomes will be examined and a transformation of the data will be used if necessary. A two-sided 5% significance level will be used for all tests without multiplicity adjustment between multiple endpoints.

#### 8.1 Sample size calculations

A sample size of 12 subjects per group has been suggested for pilot studies to evaluate feasibility and to estimate group means and standard deviations for future study planning (Julious, 2005). Based on two-sided paired t-tests and two-sample t-tests, all conducted at a 5% significance level, this pilot study will have 80% power to detect effect sizes of 0.9 for changes over time within groups and effect sizes of 1.2 for differences between groups. To account for dropout, the study will enroll 15 subjects per group, 30 total subjects.

#### 9. References

Ashina M, Goadsby PJ, Reuter U, Silberstein S, Dodick DW, Xue F, Zhang F, Paiva da Silva Lima G, Cheng S, Mikol DD. Long-term efficacy and safety of erenumab in migraine prevention: Results from a 5-year, open-label treatment phase of a randomized clinical trial. Eur J Neurol. 2021 May;28(5):1716-1725. doi: 10.1111/ene.14715. Epub 2021 Jan 20. PMID: 33400330; PMCID: PMC8248354.

de Leeuw, R, Editor, Orofacial Pain: Guidelines for Assessment, Diagnosis, and Management, The American Academy of Orofacial Pain, Sixth Edition, Hanover Park, IL: Quintessence Publishing Co, Inc., 2018, 1-25.

Edvinsson L, The CGRP Pathway in Migraine as a Viable Target for Therapies. Headache 2018;58:33-47.

Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. A controlled trial of erenumab for episodic migraine. N Engl J Med. 2017;377(22):2123–2132.

Hargreaves R, Olesen J. Calcitonin Gene-Related Peptide Modulators - The History and Renaissance of a New Migraine Drug Class. Headache 2019;59(6):951-970. doi: 10.1111/head.13510.

https://www.nidcr.nih.gov/research/data-statistics/facial-pain, July 2018.

https://www.accessdata.fda.gov/drugsatfda docs/label/2020/761077s007lbl.pdf

Headache Classification Committee of the International Headache Society (IHS), The International Classification of Headache Disorders, 3<sup>rd</sup> edition. Cephalalgia 2018;38(1): 1-211. doi: 10.1177/0333102417738202. PMID: 29368949.

Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical statistics. 2005;4:287-291.

Kean J, Monahan PO, Kroenke K, Wu J, Yu Z, Stump TE, Krebs EE. Comparative Responsiveness of the PROMIS Pain Interference Short Forms, Brief Pain Inventory, PEG, and SF-36 Bodily Pain Subscale. Med Care. 2016 Apr;54(4):414-21. doi: 10.1097/MLR.0000000000000497.

Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch S, Kroenke K. (2009). Development and Initial Validation of the PEG, a Three-item Scale Assessing Pain Intensity and Interference. Journal of General Internal Medicine, 24(6), 733–738. http://doi.org/10.1007/s11606-009-0981-1

Kroenke K, Evans E, Weitlauf S, McCalley S, Porter B, Williams T, Baye F, Lourens SG, Matthias MS, Bair MJ. Comprehensive vs. Assisted Management of Mood & Pain Symptoms (CAMMPS) trial: study design and sample characteristics. Contemporary Clin Trials 2018;64:179-187.

Kroenke K, Krebs EE, Turk D, Von Korff M, Bair MJ, Allen KD, Sandbrink F, Cheville AL, DeBar L, Lorenz KA, Kerns RD. Core outcome measures for chronic musculoskeletal pain research: recommendations from a Veterans Health Administration work group. Pain Med 2019;20(8):1500-1508.

Kroenke K, Spitzer RL, Williams JBW, Löwe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4 Psychosomatics 2009;50:613-621.

Maixner W, Fillingim RB, Williams DA, Smith SB, Slade GD. Overlapping Chronic Pain Conditions: Implications for Diagnosis and Classification. J Pain. 2016 Sep;17(9 Suppl):T93-T107. doi: 10.1016/j.jpain.2016.06.002.

Noseda R, Burstein R. Migraine pathophysiology: Anatomy of the trigeminovascular pathway and associated neurological symptoms, CSD, sensitization and modulation of pain. Pain. 2013;154(Suppl. 1):S44-S53.

Ohrbach, R, editor. Diagnostic Criteria for Temporomandibular Disorders Assessment Instruments. Version 15May2016. www.rdc-tmdinternational.org Accessed on 23Sep2019

Ohrbach R, Granger C, List T, Dworkin S. Preliminary development and validation of the Jaw Functional Limitation Scale. Community Dent Oral Epidemiol. 2008 Jun;36(3):228-36. doi: 10.1111/j.1600-0528.2007.00397.x.

Popko L. Some notes on papyrus ebers, ancient egyptian treatments of migraine, and a crocodile on the patient's head. Bull Hist Med. 2018;92(2):352-366

Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network\* and Orofacial Pain Special Interest Group. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151.

Speciali JG. Temporomandibular Dysfunction and Headache Disorder. Headache 2015;55;S1:72-83.

Tepper SJ. History and Review of anti-Calcitonin Gene-Related Peptide (CGRP) Therapies: From Translational Research to Treatment. Headache 2018;58:238-275. doi: 10.1111/head.13379.

Tepper S, Ashina M, Reuter U, et al. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017;16(6):425–434.

Toussaint A, Kroenke K, Baye F, Lourens S. Comparing the Patient Health Questionnaire - 15 and the Somatic Symptom Scale - 8 as measures of somatic symptom burden. J Psychosom Res. 2017 Oct;101:44-50. doi: 10.1016/j.jpsychores.2017.08.002.

Yuan H, Spare NM, Silberstein SD. Targeting CGRP for the Prevention of Migraine and Cluster Headache: A Narrative Review. Headache. 2019 Jul;59 Suppl 2:20-32. doi: 10.1111/head.13583.

# 10. Appendices

### **Appendix A – TMD Symptoms**

# **Symptoms of TMD:**

Jaw pain

Headache

Earache

Joint noise

Limited range of motion

Neck pain

Toothache

Shoulder pain

Dizziness

Changing bite

Ringing in the ear

Nausea

TemporoMandibular Joint pain

Locked shut

Locked open

Light sensitivity

Sound sensitivity

Hyper-sensitive facial skin

Hyper-sensitive oral mucosa

Sinus pain

Arm pain

Chest pain

(TMD symptoms mask, mimic and distort other diagnoses.)

#### Appendix B – TMD Treatments

### **Multiple types of Orthotic appliances**

Hard acrylic
Soft vinyl
Accentuated posterior stop
Accentuated anterior stop
Boil and Bite

#### **Multiple types of Occlusal rehabilitation**

Full mouth reconstruction Occlusal adjustment(s) Orthodontics

#### Multiple types of medicinal regimen

Muscle relaxants Over-the-counter NSAIDS Amitriptyline Sumatriptan

#### Multiple types of injections

TM joint injections – intracapsular diagnostic/therapeutic injections Injections of anesthetic agents into the trigeminal nerve Trigger point injections

Botulinum toxin (type A or Type B) injections

### Multiple types of surgical treatments

Alloplastic joint implants

Arthrocentesis

Arthroscopic surgery

Arthrotomy or arthroplasty

Condylectomy (partial or complete)

Disc repair procedures

Diskectomy without or with replacement

Eminectomy or eminoplasty (articular surface recontouring)

Mandibular condylotomy

Nerve obliteration

Orthognathic surgery – for correction of jaw deformities could also be done as an adjunct to definitive joint treatment when related to deformities resulting in TMJ dysfunction.

Partial or total joint reconstruction

Removal of failed implants

#### **Multiple types of Behavior Modification**

ABA

Cognitive behavior therapy Educational behavior therapy Positive Mental Attitude

#### **Other Miscellaneous Treatments**

Acupuncture

Acupressure
Allergy Treatments
Biofeedback
Chiropractic treatments
Continuous Passive Motion (CPM) therapy
Dry needling
Low level laser
Massage Therapies
Nutrition
Physical Therapy Treatments
Pulsed radiofrequency energy – Energex
Tru-Denta combination of therapies
Ultrasonic therapy with(out) medicines

### **Alternative Therapies**

Crystals
Magnets
Power bands
Pressure point bands
Tragus piercing

(Multiple non-predictable treatments suggest no predictable treatment for TMD has been found.)

#### Questionnaire Patient name Date\_ PAIN 1. Have you ever had pain in your jaw, temple, in the ear, or in front of the ear on either No Yes If you answered NO, then skip to Question 5. 2. How many years or months ago did your pain in the jaw, temple, in the months \_years ear, or in front of the ear first begin? 3. In the last 30 days, which of the following best describes No pain any pain in your jaw, temple, in the ear, or in front of the ear on either side? Pain comes and goes Select ONE response. Pain is always present If you answered NO to Question 3, then skip to Question 5. 4. In the last 30 days, did the following activities change any pain (that is, make it better or make it worse) in your jaw, temple, in the ear, or in front of the ear on either side? No Yes Chewing hard or tough food В. Opening your mouth, or moving your jaw forward or to the side C. Jaw habits such as holding teeth together, clenching/grinding teeth, or chewing D. Other jaw activities such as talking, kissing, or yawning HEADACHE 5. In the last 30 days, have you had any headaches that included the temple areas of No Yes your head? If you answered NO to Question 5, then skip to Question 8. 6. How many years or months ago did your temple headache first begin? vears months 7. In the last 30 days, did the following activities change any headache (that is, make it better or make it worse) in your temple area on either side? Nο Yes Chewing hard or tough food A. В. Opening your mouth, or moving your jaw forward or to the side Jaw habits such as holding teeth together, clenching/grinding, or chewing gum C. Other jaw activities such as talking, kissing, or yawning D

Appendix C - Diagnostic Criteria for Temporomandibular Disorders Symptom

Copyright International RDC/TMD Consortium Network. Available at <a href="http://www.rdc-tmdinternational.org">http://www.rdc-tmdinternational.org</a> Version 12May2013. No permission required to reproduce, translate, display, or distribute.

| JAV | W JOINT NOISES | | | Office u | ıse |
|---|---|---|---|---|---|
| 8. | In the last 30 days, have you had any jaw joint noise(s) when you moved or used your jaw? | No | Yes | R L | DNK |
| CLO | OSED LOCKING OF THE JAW | | - | | |
| 9. | Have you <u>ever</u> had your jaw lock or catch, even for a moment, so that it would <u>not open</u> ALL THE WAY? | | | | |
| | If you answered NO to Question 9 then skip to Question 13. | | | | |
| 10. | Was your jaw lock or catch severe enough to limit your jaw opening and interfere with your ability to eat? | | | | |
| 11. | In the last 30 days, did your jaw lock so you could <u>not open</u> ALL THE WAY, even for a moment, and then unlock so you could open ALL THE WAY? | | | | |
| | If you answered NO to Question 11 then skip to Question 13. | | | | |
| 12. | Is your jaw currently locked or limited so that your jaw will <u>not open</u> ALL THE WAY? | | | | |
| ОР | EN LOCKING OF THE JAW | | | | |
| 13. | In the last 30 days, when you opened your mouth wide, did your jaw lock or catch even for a moment such that you could <u>not close</u> it from this wide open position? | | | | 10 - |
| | If you answered NO to Question 13 then you are finished. | | | The second secon | |
| 14. | In the last 30 days, when you jaw locked or caught wide open, did you have to do something to get it to close including resting, moving, pushing, or maneuvering it? | | | | |

Copyright International RDC/TMD Consortium Network. Available at <a href="http://www.rdc-tmdinternational.org">http://www.rdc-tmdinternational.org</a> Version 12May2013. No permission required to reproduce, translate, display, or distribute.

# Appendix D – Brief Pain Inventory (BPI)

# **BRIEF PAIN INVENTORY (BPI)**

For the following questions, please answer for your facial, jaw or TMD pain:

| the lor | lowing | questic | ms, pre | ase ans | wei iui | your 1 | aciai, ja | IW OI I | MID pa | 1111. | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | nse rate<br>ne last v | | ain by c | ircling t | he one 1 | number | that bes | st descri | bes you | ur pain at | its <u>worst</u> |
| 0<br>No<br>Pain | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | ] | 10<br>Pain as ba<br>1 can ima | |
| | nse rate<br>ne last v | - | nin by c | ircling t | he one 1 | number | that bes | st descri | bes you | ur pain at | its <u>least</u> |
| 0<br>No<br>Pain | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | ] | 10<br>Pain as ba<br>a can ima | |
| | ise rate<br><u>rage</u> . | your pa | nin by c | ircling t | he one 1 | number | that bes | st descri | bes you | ur pain oi | n the |
| 0<br>No<br>Pain | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | ] | 10<br>Pain as ba<br>1 can ima | |
| 4. Plea | | your pa | nin by c | ircling t | he one 1 | number | that tell | ls how 1 | nuch p | ain you h | ave <u>right</u> |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |

Circle the number that describes how, during the past week, pain has interfered with your:

0 1 2 3 4 5 6 7 8 9 10

Does Not

Interfere

Interferes

5. General Activity

No Pain Pain as bad as

you can imagine

| 6. Mood | 1 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 0<br>Does Not<br>Interfere | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| 7. Walk | ing Abi | ility | | | | | | | | |
| 0<br>Does Not<br>Interfere | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| 8. Norm | 8. Normal Work (includes both work outside the and housework) | | | | | | | | | |
| 0<br>Does Not<br>Interfere | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| 9. Relat | ions wi | th other | People | | | | | | | |
| 0<br>Does Not<br>Interfere | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| 10. Sleep | , | | | | | | | | | |
| 0<br>Does Not<br>Interfere | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| 11. Enjoy | ment o | f Life | | | | | | | | |
| 0<br>Does Not<br>Interfere | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |

# Appendix E - PEG (Pain, Enjoyment, General Activity) Scale and Pain Medication Assessment

# **PEG Pain**

| For the following questions | , please answer for | your facial, jaw o | or TMD pain: |
|---|---|---|---|
|---|---|---|---|

| | | | | | | _ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1. | What nu | ımber | best de | escribes | s your | pain o | n the <u>a</u> | <u>verage</u> | in the | last 24 | 1 hours? | |
| | 0<br>No<br>Pain | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>iin as bad as<br>can imagine | |
| 2. | What nu | | | escribes | s how, | , in the | last 24 | hours, | pain h | nas inte | erfered with | your |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | es Not<br>nterfere | | | | | | | | | | Completely<br>Interferes | |
| 3. | What nu | | | escribes | s how, | , in the | last 24 | hours, | pain h | nas inte | erfered with | your |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | es Not<br>nterfere | | | | | | | | | | Completely<br>Interferes | |

# **Pain Medication Assessment Questions**

- A. Did you take any medicines for pain today?
  - Yes
  - No
- B. If YES, were any of these medicines you took today for facial, jaw or TMD pain?
  - Yes
  - No

# **Appendix F – Patient Global Impression of Change (PGIC)**

# Patient Global Impression of Change (PGIC)

Since the start of the study (treatment), my overall facial, jaw or TMD pain is ....

- 1. Much better
- 2. Moderately better
- 3. A little better
- 4. No change
- 5. A little worse
- 6. Moderately worse
- 7. Much worse

Version Date: Amend 8- January 12, 2023 Page 23 of 27

### **Appendix G – Jaw Function Limitation Scale (JFLS-8)**

# **Jaw Functional Limitation Scale - 8**

For each of the items below, please indicate the level of limitation **during the last month.** If the activity has been completely avoided because it is too difficult, then circle '10'. If you avoid an activity for reasons other than pain or difficulty, leave the item blank.

| | No<br>Limit | atio | n | | | | | | | | evere<br>mitation |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1. Chew tough food | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 2. Chew chicken (e.g., prepared in oven) | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 3. Eat soft food requiring no chewing (e.g., mashed potatoes, apple sauce, pudding, pureed food) | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 4. Open wide enough to drink from a cup | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 5. Swallow | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 6. Yawn | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 7. Talk | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 8. Smile | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |

Copyright Ohrbach R. Available at <a href="http://www.rdc-tmdinternational.org">http://www.rdc-tmdinternational.org</a>
Version 12May2013. No permission required to reproduce, translate, display, or distribute.

# Appendix H – Depressive and anxiety symptoms (PHQ-4)

# PHQ-4: Depression (PHQ-2) and Anxiety (GAD-2)

| b | r the <u>last 2 weeks</u> , how often have you been othered by any of the following problems? | Not at<br>all | Several<br>days | More than half the days | Nearly<br>every<br>day |
|---|---|---|---|---|---|
| Use a check (✓) to indicate your answer for each item | | (0) | (1) | (2) | (3) |
| 1. | Feeling nervous anxiety or on edge | | | | |
| 2. | Not being able to stop or control worrying | | | | |
| 3. | Little interest or pleasure in doing things | | | | |
| 4. | Feeling down, depressed, or hopeless | | | | |

Version Date: Amend 8- January 12, 2023 Page 25 of 27

# Appendix I – Somatic symptom severity as measured by the SSS-8

# **Somatic Symptom Scale (SSS-8)**

# During the <u>past 7 days</u>, how much have you been bothered by any of the following problems?

| | Not<br>at all | A little<br>bit | Some what | Quite a<br>bit | Very<br>much |
|---|---|---|---|---|---|
| 1. Stomach or bowel problems | <u> </u> | 1 | _ 2 | □ 3 | 4 |
| 2. Back pain | □ 0 | 1 | _ 2 | □ 3 | 4 |
| 3. Pain in your arms, legs, or joints | □ 0 | 1 | <u> </u> | □ 3 | <u> </u> |
| 4. Headaches | □ 0 | 1 | _ 2 | □ 3 | 4 |
| 5. Chest pain or shortness of breath | □ 0 | 1 | _ 2 | □ 3 | 4 |
| 6. Dizziness | □ 0 | 1 | <u> </u> | □ 3 | <u> </u> |
| 7. Feeling tired or having low energy | □ 0 | <u> </u> | <u> </u> | □ 3 | <u> </u> |
| 8. Trouble sleeping | □ 0 | 1 | <u> </u> | □ 3 | <u> </u> |

#### 11. Table 1

# ISS – Timeframes for Submission of Safety Data to Amgen

For Interventional studies with Amgen IMPa:

| Safety Data | Timeframe for submission to Amgen | Send to |
|---|---|---|
| Suspected Unexpected Serious | At time of regulatory submission | Amgen Safety |
| Adverse Reaction (SUSARs) | | |
| Pregnancy/Lactation exposure and any associated reports/outcomes (i.e. unexpected pregnancy, pregnancy of partner, spontaneous abortion, congenital anomaly etc.) | Within 1 business day of Sponsor<br>awareness, for reports meeting serious<br>criteria<br>Not to exceed 15 calendar days of Sponsor<br>awareness, for non-serious reports | Amgen Safety |

<sup>&</sup>lt;sup>a</sup> Specific requirements are to be outlined in the Research Agreement.

For all study types – aggregate reports<sup>a</sup>(as applicable):

| Safety Data | Timeframe for submission to Amgen | Send to |
|---|---|---|
| Listing for Safety data | Once per year and at the end of the | NASCR Manager |
| reconciliation <sup>b</sup> | study | |
| Annual Safety Report | | |
| (eg, EU Clinical Trial Directive | Annually | NASCR Manager |
| DSUR and US IND Annual | | |
| Report) | | |
| Other aggregate analyses | At the time of Sponsor submission to any | NASCR Manager |
| (any report containing Safety data | body governing research conduct (eg. | |
| generated during the course of | RA, IRB etc.) | |
| the study) | | |
| Final (End of Study Report, | | |
| including): | At the time of Sponsor submission to any | NASCR Manager |
| <ul> <li>Unblinding data for</li> </ul> | body governing research conduct (eg. | |
| blinded studies | RA, IRB etc.) but no later than 1 calendar | |
| <ul> <li>Reports of unauthorized</li> </ul> | year of study completion | |
| use of a marketed product | | |

<sup>&</sup>lt;sup>a</sup> Specific requirements are to be outlined in the Research Agreement.

<sup>&</sup>lt;sup>b</sup> Listing for reconciliation should include all ICSRs submitted to Amgen Safety per contract (i.e. for studies in Table 1 listing should include ADRs, SADRs, Other Safety Findings, USADEs, SADEs and non-serious ADEs; for studies in Table 2 listing should contain SUSARs, pregnancy and lactation exposure (and any associated reports/outcomes), USADEs, SADEs and non-serious ADEs; studies in table 3 do not require reconciliation).